CLINICAL TRIAL: NCT03249415
Title: Endometrial Reconstruction by Human Regenerative Factors Derived From Platelet-Rich Plasma in Mice Models
Brief Title: Use of PRP in Endometrial Reconstruction
Status: Completed | Type: Observational
Sponsor: Fundación IVI (Other)
Responsible Party: Sponsor
Other Study IDs: 1701-FIVI-003-IC
Record Dates: First submitted 2017-06-08; First posted 2017-08-15 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Asherman Syndrome; Endometrial Atrophy
Keywords: Platelet-Rich Plasma; Cell therapy; Regenerative factors; Autologous treatment; Paracrine factors
MeSH Terms: conditions — Gynatresia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Platelet-Rich Plasma from Whole Blood.

SUMMARY:
Infertility, which affected 48.5 million couples worldwide in 2010 alone, has many causes; some causes result from issues related to the endometrium. Unfortunately, no cure exists for medical conditions resulting in the destruction of the endometrium, or for non-functional uterus. Thus, safe and effective therapies are needed to treat these diseases and to establish fertility in affected women. These novel techniques refer to the use and application of regenerative/paracrine factors to regenerate the endometrium in patients with Asherman's Syndrome (AS) and Endometrial Atrophy (EA).These new therapies based on the injection of the identified regenerative/paracrine factors and the platelet-rich plasma (PRP) from whole blood in an immunodeficient mouse model with AS/EA, evaluating their contribution and/or effect in the endometrial repair by functional proofs.

DETAILED DESCRIPTION:
The objective is to know the effect of these regenerative factors obtained from Platelet-Rich Plasma in an immunodeficient murine model with AS/EA Blood from patients with Asherman's Syndrome (AS) and Endometrial Atrophy (EA) will be collected, maintained under anticoagulant solution and after several centrifugations PRP will be obtained. Demonstration of a functional endometrium will be proved determining pregnancy and implantation rates as well as the number of live pups/pregnant female in our mice model. Also, the uterus histology will be analysed in treated and untreated mice

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with Asherman Syndrome and Endometrial Atrophy by Hysteroscopy.
* No pregnancy after hormonal treatment.

Exclusion Criteria:

* Psychiatric diseases.

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Participant with endometrial pathologies.
Study Population: Participants diagnosed with Asherman Syndrome and Endometrial Atrophy by Hysteroscopy.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-07-18 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Endometrial thickness after reconstruction in murine model | through study completion, an average of 1 year
  Using histological and functional technologies demonstration of regeneration ability of PRP

CONTACTS AND LOCATIONS:
Overall Officials: Irene Cervello, PhD, Principal Investigator — Fundación IVI
Locations (1):
- IVI Barcelona, Barcelona, Spain

REFERENCES:
- [Result] Cervello I, Gil-Sanchis C, Santamaria X, Cabanillas S, Diaz A, Faus A, Pellicer A, Simon C. Human CD133(+) bone marrow-derived stem cells promote endometrial proliferation in a murine model of Asherman syndrome. Fertil Steril. 2015 Dec;104(6):1552-60.e1-3. doi: 10.1016/j.fertnstert.2015.08.032. Epub 2015 Sep 15. PMID 26384164